CLINICAL TRIAL: NCT01843868
Title: A Single Arm Study to Evaluate the Control of Chemotherapy Induced Nausea and Vomiting in Non-Hodgkin Lymphoma Patients Receiving R-CHOP.
Brief Title: Emesis Control Study in Non-Hodgkin Lymphoma Patients Receiving R-CHOP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant due to protracted logistical and subsequent funding matters.
Sponsor: Australasian Leukaemia and Lymphoma Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ALLG SC03; ACTRN12611001269921 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2013-04-24; First posted 2013-05-01 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphoma; Non-Hodgkin; Emesis; Chemotherapy; Nausea; Vomiting; Aprepitant
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Vomiting; Nausea | interventions — R-CHOP protocol; Rituximab; Doxorubicin; Vincristine; Cyclophosphamide; Prednisolone; Antiemetics; Ondansetron; Granisetron; Tropisetron; Palonosetron; Metoclopramide; Prochlorperazine; Lorazepam; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOP and standard anti-emetics (Other): This is a single arm study.
  All patients receive R-CHOP every 14 or 21 days for a minimum of 3 cycles. Standard anti-emetics will be used as follows:
  * 5HT3 (5-Hydroxytryptamine 3) antagonists (ondansetron, granisetron or tropisetron) used as the local institutional standard of care will be permitted, although the preferential use of ondansetron or granisetron will be encouraged.
  * Dexamethasone will not to be used as patients receive hydrocortisone and oral prednisolone in R-CHOP. In this study, the use of oral prednisolone on day 1 will be regarded as equivalent to dexamethasone. Prednisolone will be given PRIOR to the chemotherapy with the 5HT3 antagonist.
  * Anti-emetics (metoclopramide, prochlorperazine and lorazepam) may be prescribed to be used 'as needed' for breakthrough emesis.
  * Patients 'failing' the standard Chemotherapy Induced Nausea and Vomiting prophylactic regimen will be eligible to receive aprepitant (Days 1 to 3) for subsequent cycles.
  Interventions: Drug: Standard anti-emetics in conjunction with R-CHOP

INTERVENTIONS:
Drug: Standard anti-emetics in conjunction with R-CHOP
  Other Names: R-CHOP:; rituximab; doxorubicin; vincristine; cyclophosphamide; prednisolone; Anti-emetics:; ondansetron; granisetron; tropisetron; palonosetron; metoclopramide; prochlorperazine; lorazepam; aprepitant

SUMMARY:
The incidence and severity of chemotherapy-induced nausea and vomiting (CINV) in patients receiving R-CHOP chemotherapy for in non-Hodgkin's lymphoma is not well documented. The contribution of prednisolone to CINV control in the R-CHOP regimen is also unclear.

This study aims to evaluate the overall effectiveness of antiemetic control using a standardised 5HT3 (5-Hydroxytryptamine 3) antagonist-containing regimen (e.g. ondansetron) in a heterogeneous group of patients receiving R-CHOP chemotherapy (Rituximab Doxorubicin Vincristine Cyclophosphamide Prednisolone).

DETAILED DESCRIPTION:
The aim of this study will be to investigate the incidence and severity of CINV in patients receiving R-CHOP for the treatment of non-Hodgkin lymphoma and standardised antiemetic prophylaxis.

The study hypothesises that the control of delayed nausea and emesis is suboptimal in a proportion of patients receiving R-CHOP regimens and that delayed CINV is not prevented by use of 5HT3 antagonists beyond the first day of use post-chemotherapy administration.

Participating institutions will prospectively collect data on the incidence of CINV, the severity of CINV, the use of break through/rescue medication for episodes of CINV uncontrolled by prescribed regular antiemetics, the effectiveness of additional measures used when previous CINV control has been inadequate (for example the use of aprepitant as an additional measure in subsequent cycles) and the major side-effects likely to be related to the antiemetics.

The analysis of these results will determine the incidence and severity of CINV in patients receiving R-CHOP and the effectiveness of the prescribed antiemetic regimens. Analysis will also determine if the control and incidence of CINV is a significant problem in defined subgroups of patients receiving R-CHOP and could inform the design of future research (or an extension of the current protocol) in this area. Sub groups for investigation will include patients with advanced disease, those with abdominal involvement, those receiving R-CHOP every 14 days versus every 21 days (R-CHOP14 versus R-CHOP21), those receiving 6 or 8 treatment cycles of R-CHOP, older patients, younger females etc. A potential randomised study evaluating the role of aprepitant could be contemplated in high risk groups.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of non Hodgkin's Lymphoma
2. Newly diagnosed or relapsed patients who are chemotherapy-naïve or who have not received chemotherapy in the last 12 months. Pre-phase therapy with prednisolone and/or vincristine for < one week duration prior to commencement of cycle 1 of R-CHOP is permissible
3. Intended to receive R-CHOP every 14 or 21 days for minimum 3 cycles with rituximab planned to be given with CHOP on day 1 or fractionated over days 1 and 21.
4. Males and females, age 18 years or older
5. Are reasonably expected to be able to complete the CINV tool
6. Willing to complete assessments and tool as required for the study
7. ECOG (Eastern Cooperative Oncology Group) performance status score of 2 or less
8. Has provided written informed consent

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Previous adverse reaction to the standard anti-emetics proposed in the study
3. Contraindications to the use of the anti-emetics included as standard of care in the study (e.g. cardiac, liver function)
4. Participation in other therapeutic studies investigating CINV.
5. Has any other clinically important abnormalities as determined by the investigator that may interfere with his or her participation in or compliance with the study
6. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01 (Estimated); Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Complete Response, Acute Phase (Day 1), Cycle 1 | Day 1
  The proportion of patients experiencing a complete response defined as no vomiting and no use of breakthrough medication in the acute phase (day 1: 0 - 24 hours) of the first cycle of R-CHOP chemotherapy
Complete Response, Delayed Phase (Days 2 to 11), Cycle 1 | Days 2 to 11
  The proportion of patients experiencing a complete response defined as no vomiting and no use of breakthrough medication in the delayed phase (days 2 - 11 inclusive) of the first cycle of R-CHOP chemotherapy

SECONDARY OUTCOMES:
Complete Response - Cycle 2 and beyond | Day 1 to Day 11
  Complete response in the acute and delayed phases of each of cycles 2 and beyond of R-CHOP chemotherapy
No Significant Nausea - Cycle 2 and beyond | Day 1 to Day 11
  No significant nausea (defined as a nausea experience score of <2.5cm on a 0 - 10cm visual analogue scale) in the acute and delayed phases of each of cycles 2 and beyond of R-CHOP chemotherapy
Failure of standard anti-emetic prophylaxis, Day 1 to Day 11, Cycle 1 and beyond | Day 1 to Day 11
  Failure of standard anti-emetic prophylaxis in the acute and delayed phase of any one cycle of chemotherapy requiring aprepitant as secondary prophylaxis in subsequent cycles. Failure will be defined as the occurrence of any of the following either during or beyond cycle day 1:
  * One or more episodes of vomiting
  * One or more episodes of nausea requiring the use of 1 or more doses of breakthrough anti-emetics
  * An episode of nausea requiring the use of breakthrough anti-emetics across multiple days
  * An episode of nausea measuring > 2.5cm on a 0 - 10cm visual analogue scale
  * Nausea and/or vomiting that in the clinicians opinion requires use of aprepitant in future cycles
Frequency of common adverse events associated with anti-emetics | Day 1 to Day 11
  Adverse Events (all grades) of the anti-emetic regimen in each cycle of R-CHOP chemotherapy
Severity of common adverse events associated with anti-emetics | Day 1 to Day 11
  Adverse Events (all grades) of the anti-emetic regimen in each cycle of R-CHOP chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Grigg, Professor, Principal Investigator — Director of Clinical Haematology, Austin Hospital, Australia